CLINICAL TRIAL: NCT00802750
Title: A Randomized, Single-blind, Cross-over, Single Centre Study in Healthy Volunteers Evaluating Subject Perception of Urinary Catheters Manufactured in a New Process With New Solvent
Brief Title: Study Where Healthy Volunteers Evaluate LoFric Catheters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wellspect HealthCare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: YA-LSM-0001
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Catheterization

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Device: LoFric POBE
- B (Experimental)
  Interventions: Device: LoFric POBE

INTERVENTIONS:
Device: LoFric POBE — LoFric POBE, Nelaton 40 cm, CH 12 with new solvent. Each subject will use the reference catheter "LoFric POBE, Nelaton 40 cm, CH 12 with current solvent" before being catheterized with the test catheters.
  Arms: A
Device: LoFric POBE — Unsalted LoFric POBE Hydro-Kit II, Nelaton 40 cm, CH 12 with new solvent Each subject will use the reference catheter "LoFric POBE, Nelaton 40 cm, CH 12 with current solvent" before being catheterized with the test catheters.
  Arms: B

SUMMARY:
The purpose of this study is to evaluate healthy volunteers perception of catheterization with LoFric catheters with new solvents in the manufacturing process. The subjects will be catheterized three times during one visit day.

The hypothesis is that the subjects' perception of catheterization is the same when using the test catheters compared to the reference catheter.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Healthy volunteers
* Males age 18 years and over

Exclusion Criteria:

* Known or suspected, current impairment of and/or decreased urethral sensibility
* History of urethral disease
* History of urinary tract infection within three months, or ongoing symptomatic urinary tract infection
* Use of medications that may affect the urethra's dryness (e. g. anti-cholinergic drugs or cortisone)
* Current drug, alcohol or other substance abuse
* Other significant disease or condition (e.g. benign prostate hypertrophy, other prostatic lesions), which may interfere with treatment and/or evaluation
* Allergy to Trimethoprim
* Suspected poor compliance with the protocol during the complete study period.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-11; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Healthy volunteers perception of catheterization | At each catheterization (three times during one day)

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Malmqvist, MD, PhD, Assoc.Prof., Principal Investigator — Clinical Research and Trial Centre, Lund University Hospital
Locations (1):
- Clinical Research and Trial Centre, Lund University Hospital, Lund, Sweden